CLINICAL TRIAL: NCT01760512
Title: Prospective, Single-blind, Randomized, Non-inferiority, and Controlled Study of Clinical and Health Economic Impact of Robot-assisted Surgery Versus Conventional Laparoscopy in Bariatric Surgery: the Case of Gastric Bypass
Brief Title: Clinical and Health Economic Impact of Robot-assisted Surgery vs Conventional Laparoscopy : the Case of Gastric Bypass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IHU Strasbourg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12-002
Record Dates: First submitted 2012-12-10; First posted 2013-01-04 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-05

CONDITIONS: Morbid Obesity
Keywords: Gastric bypass; Robot-assisted surgery; Conventional laparoscopy; Pain assessment; Health economics outcomes
MeSH Terms: conditions — Obesity, Morbid | interventions — Gastric Bypass

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Robot-assisted surgery (Experimental): Robot-assisted (da Vinci surgical system) gastric bypass
  Interventions: Procedure: Gastric bypass
- Conventional laparoscopy (Active Comparator): Laparoscopic gastric bypass
  Interventions: Procedure: Gastric bypass

INTERVENTIONS:
Procedure: Gastric bypass — Gastric bypass

SUMMARY:
The purpose of this study is to gather clinical and economic evidence on the use of robotics for bariatric surgery (gastric bypass).

This monocentric, randomized, single blind, controlled study will evaluate post-operative pain, quality of life and appetite, post-operative complication incidence. It will also provide information on direct and indirect costs of surgery.

DETAILED DESCRIPTION:
Robot-assisted Surgery Versus Conventional Laparoscopy in Bariatric Surgery (Gastric Bypass): a prospective, single-blind, randomized, non-inferiority, and controlled study The main evaluation criterion is 24h post-operative pain assessed using visual analog scale (VAS). Secondary criteria included for clinical assessment: post 24h pain, excess weight loss, quality of life, appetite, complications, conversion rate; and for health-economics assessment : duration of surgical steps, length of stay, return to normal activity and their conversion to cost, consumables, estimation of indirect costs and benefits (e.g., robotics perception, publication).

In this study, main inclusion criteria include major obesity (IMC ≥ 35) with co-morbidities or morbid obesity (IMC ≥ 40), scheduled gastric bypass surgery Main contraindications are previous bariatric surgery and previous major abdominal surgeries To test robotic-assisted surgery non-inferiority on VAS pain score 24h post-surgery, a total of 128 patients (64 per arm) is to be included (alpha 2,5%; power 90%; drop-out rate: 5%).

The study will include 12 months of follow-up post-surgery for each patient. The total study duration is 2 years and 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient presenting with major obesity (BMI ≥ 35) with co-morbidities or morbid obesity (BMI ≥ 40)according to French HAS (Haute Autorité de Santé) and CNAMTS (Caisse nationale de l'assurance maladie des travailleurs salariés)criteria for whom gastric bypass is scheduled
* Male or female between 18 and 65 years old
* Patient registered with the French Social Security
* Patient having provided a written informed consent prior to enrolment
* Patient accepting to attend follow-up visits as required by study protocol

Exclusion Criteria:

* Patient with a BMI ≥ 60
* Patient with a contraindication for laparoscopic gastric bypass with or without robotic assistance
* Patient having had prior bariatric surgery
* Patient having had prior major abdominal surgery
* Patient in exclusion period of another clinical study
* Patient pregnant or breastfeeding
* Patient without sufficient knowledge of french language or unable to receive or understand study related information and answer to questionnaires
* Patient with no or limited legal capacity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2012-11; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
24h postoperative pain | 24h
  Pain assessment 24h post surgery (visual analog scale)

SECONDARY OUTCOMES:
Evaluation of post-operative pain | 24h, 8 days, 1, 3, 6 and 12 months
  Evaluation of post-operative pain (beyond 24h post-operative) using VAS
Evaluation of quality of life (BAROS and GIQLI) | At 1, 3, 6 and 12 months
  Evaluation of quality of life using BAROS and GIQLI questionaires
Evaluation of appetite level | At 8 days, 1, 3, 6 and 12 months
  Evaluation of appetite level using VAS
Percentage of excess weight loss | At 8 days, 1, 3, 6 and 12 months
  Measure of excess weight loss - % from baseline
Conversion rate to conventional laparoscopy | During the procedure (Day 0)
  Conversion rate to conventional laparoscopy (only applicable to robot-assisted surgery arm)
Nature of per-operative complications | During the procedure (Day 0)
  Nature of per-operative complications
Nature of post-operative complications | Following the procedure (Day 0) up to 12 months
  Nature of post-operative complications
Evaluation of operative times | During the procedure (Day 0)
  Evaluation of key steps of gastric bypass surgery, OR occupation time
Evaluation of direct costs | During the procedure (day 0) and up to 12 months
  Direct costs include material used, OR occupation time, length of stay, return to normal activity
Evaluation of indirect costs | Up to 12 months
  Combination of number of patients having surgery, perception of robot-assisted surgery by both personnel and patients, publications, and communications

CONTACTS AND LOCATIONS:
Overall Officials: Michel Vix, Principal Investigator — Service de Chirurgie Générale et Endocrinienne - Nouvel Hôpital Civil - Strasbourg
Locations (1):
- Service de Chirurgie Digestive et Endocrinienne, Strasbourg, France